CLINICAL TRIAL: NCT00452023
Title: PEG IFN-alpha2a (Pegasys®) Therapy in Patients With Chronic Myeloproliferative Diseases (Excluding Philadelphia Chromosome Positive Chronic Myeloid Leukemia)
Brief Title: Pegasys® in Patients With Myeloproliferative Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM03-0109; NCI-2012-01474 (Registry Identifier: NCI CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2007-03-22; First posted 2007-03-26 (Estimated); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Myeloproliferative Disorders
Keywords: Myeloproliferative Disorders; Essential Thrombocythemia; Polycythemia Vera; Pegasys; IFN-alpha2a; Pegylated-Interferon Alpha-2A; PEG-IFNa-2a
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombocythemia, Essential; Polycythemia Vera | interventions — Interferon alpha-2; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- IFN-alpha2a 90 Microgram (mcg) weekly (Experimental): Starting dose 90 microgram (mcg) injection under the skin once a week.
  Interventions: Drug: IFN-alpha2a
- IFN-alpha2a 450 Microgram (mcg) weekly (Experimental): Starting dose 450 microgram (mcg) injection under the skin once a week.
  Interventions: Drug: IFN-alpha2a
- IFN-alpha2a 360 Microgram (mcg) weekly (Experimental): Starting dose 360 microgram (mcg) injection under the skin once a week.
  Interventions: Drug: IFN-alpha2a
- IFN-alpha2a 270 Microgram (mcg) weekly (Experimental): Starting dose 270 microgram (mcg) injection under the skin once a week.
  Interventions: Drug: IFN-alpha2a
- IFN-alpha2a 180 Microgram (mcg) weekly (Experimental): Starting dose 180 microgram (mcg) injection under the skin once a week.
  Interventions: Drug: IFN-alpha2a

INTERVENTIONS:
Drug: IFN-alpha2a — Starting dose 90 microgram (mcg) injection under the skin once a week
  Other Names: Pegylated-Interferon Alpha-2A; PEG-IFNa-2a; Pegasys

SUMMARY:
The goal of this clinical research study is to see if Pegasys (IFN-alpha2a) can help to control the disease in patients with ET, PV, AMM/MF, and Ph-negative CML. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
IFN-alpha2a has been used for the treatment of a variety of disorders (such as hepatitis C). IFN-alpha2a is a drug that may affect the way infections and malignant diseases develop.

Before treatment starts, you will have blood (around 2 teaspoons) and bone marrow samples collected. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. These samples will be used for tests to confirm the diagnosis of the disease. Women who are able to have children must have a negative blood pregnancy test.

During treatment, you will receive IFN-alpha2a as an injection under the skin once a week. You (or your caregiver) will be taught how to give the injections, and you will receive treatment on an outpatient basis.

Treatment will continue (injections once a week) as long as the disease does not get worse.

If the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

During treatment you will have blood (around 1 teaspoon) collected every other week for 2 months, then once every 1 or 2 months for a year, then every 3 months. You will also have bone marrow samples collected every 3 to 6 months during the first year of treatment. After the first year of treatment, bone marrow samples will be collected only when your doctor feels they are needed. The blood and bone marrow samples will be used for tests to check on the response to therapy.

This is an investigational study. IFN-alpha2a has been approved by the FDA for the treatment of hepatitis C and is commercially available. However the use of IFN-alpha2a in this study is investigational. The commercial prepartion of IFN-alpha2a(Pegasys) will be used in this study. Up to 280 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Following diagnoses: --ET: Patients with PLT > 600 x10 9 /l documented in the past 12 months; hyperplasia of marrow megakaryocytes in the absence of identifiable cause of thrombocytosis and in the absence of Ph chromosome. Patients with ET and lower PLT will be eligible if attributable to prior ET therapy. --PV: Patients should have Hb >/= 15g/dl (except if patient is having phlebotomies done) and documented past diagnosis.
2. Performance status </= 2 (ECOG scale).
3. Age greater than 18 years since disease is extremely rare in younger age group.
4. Adequate liver function: total bilirubin of </= 2.0 mg/dl (except for patients with Gilbert's Syndrome) and AST (SGOT) or ALT (SGPT) < 3 X ULN (or < 5 X ULN if considered due to tumor), and renal function (serum creatinine </= 2.0 mg/dl).
5. Signed informed consent indicating that patients are aware of the investigational nature of this study in keeping with the policies of the M.D. Anderson Cancer Center. The only acceptable consent form is the one approved by the M.D. Anderson Cancer Center IRB.
6. Willingness and ability to comply with the requirements of the protocol for the duration of the study.
7. Patients must have been off chemotherapy for 1 week prior to beginning Pegasys and have recovered from the toxic effects of that therapy. Patients may have received hydroxyurea or anagrelide immediately before study entry, and may continue into therapy if treating physician determines this is in the best interest of the patient.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with prior history of another malignancy or concurrent malignancy, except for the following: basal cell carcinoma of the skin, carcinoma in situ of the cervix, or other malignancies if the patient is disease free >3 years.
3. Patients with history of ischemic retinopathy.
4. Patients with history of severe cardiac disease: NYHA Functional Class III or IV, myocardial infarction within 6 months, uncontrolled ventricular tachyarrhythmias or unstable angina.
5. Patients with history of medically significant psychiatric disease if not controlled, especially endogenous depression (does not include reactive depression post-cancer diagnosis), psychosis and bipolar disease.
6. Patients with seizure disorders requiring anticonvulsant therapy.
7. Patients with known infection with HBV, HIV, or other active systemic infection.
8. Patients with known autoimmune disease except for rheumatoid arthritis.
9. Patients with renal disease on hemodialysis.
10. Patients taking continuous or chronic high-dose systemic steroids; if discontinued, there must be a minimum washout period of one month before study drug is begun.
11. Patients with known hypersensitivity to PEG-IFN alpha-2a or its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-04-07 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Masarova, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Masarova L, Yin CC, Cortes JE, Konopleva M, Borthakur G, Newberry KJ, Kantarjian HM, Bueso-Ramos CE, Verstovsek S. Histomorphological responses after therapy with pegylated interferon alpha-2a in patients with essential thrombocythemia (ET) and polycythemia vera (PV). Exp Hematol Oncol. 2017 Nov 9;6:30. doi: 10.1186/s40164-017-0090-5. eCollection 2017. PMID 29152412
- [Derived] Masarova L, Patel KP, Newberry KJ, Cortes J, Borthakur G, Konopleva M, Estrov Z, Kantarjian H, Verstovsek S. Pegylated interferon alfa-2a in patients with essential thrombocythaemia or polycythaemia vera: a post-hoc, median 83 month follow-up of an open-label, phase 2 trial. Lancet Haematol. 2017 Apr;4(4):e165-e175. doi: 10.1016/S2352-3026(17)30030-3. Epub 2017 Mar 11. PMID 28291640
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- IFN-alpha2a 450 Microgram (mcg) Injection: Starting dose 450 microgram (mcg) injection under the skin once a week.
  IFN-alpha2a: Starting dose 450 microgram (mcg) injection under the skin once a week
- IFN-alpha2a 360 Microgram (mcg) Injection: Starting dose 360 microgram (mcg) injection under the skin once a week.
  IFN-alpha2a: Starting dose 360 microgram (mcg) injection under the skin once a week
- IFN-alpha2a 270 Microgram (mcg) Injection: Starting dose 270 microgram (mcg) injection under the skin once a week.
  IFN-alpha2a: Starting dose 270 microgram (mcg) injection under the skin once a week
- IFN-alpha2a 180 Microgram (mcg) Injection: Starting dose 180 microgram (mcg) injection under the skin once a week.
  IFN-alpha2a: Starting dose 180 microgram (mcg) injection under the skin once a week
- IFN-alpha2a 90 Microgram (mcg) Injection: Starting dose 90 microgram (mcg) injection under the skin once a week.
  IFN-alpha2a: Starting dose 90 microgram (mcg) injection under the skin once a week
Period: Overall Study
Arm/Group | IFN-alpha2a 450 Microgram (mcg) Injection | IFN-alpha2a 360 Microgram (mcg) Injection | IFN-alpha2a 270 Microgram (mcg) Injection | IFN-alpha2a 180 Microgram (mcg) Injection | IFN-alpha2a 90 Microgram (mcg) Injection
Started | 3 | 3 | 19 | 26 | 32
Completed | 3 | 3 | 19 | 26 | 32
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- IFN-alpha2a 450 Microgram (mcg): Starting dose 450 microgram (mcg) injection under the skin once a week.
  IFN-alpha2a: Starting dose 450 microgram (mcg) injection under the skin once a week
- IFN-alpha2a 360 Microgram (mcg): Starting dose 360 microgram (mcg) injection under the skin once a week.
  IFN-alpha2a: Starting dose 360 microgram (mcg) injection under the skin once a week
- IFN-alpha2a 270 Microgram (mcg): Starting dose 270 microgram (mcg) injection under the skin once a week.
  IFN-alpha2a: Starting dose 270 microgram (mcg) injection under the skin once a week
- IFN-alpha2a 180 Microgram (mcg): Starting dose 180 microgram (mcg) injection under the skin once a week.
  IFN-alpha2a: Starting dose 180 microgram (mcg) injection under the skin once a week
- IFN-alpha2a 90 Microgram (mcg): Starting dose 90 microgram (mcg) injection under the skin once a week.
  IFN-alpha2a: Starting dose 90 microgram (mcg) injection under the skin once a week
- Total: Total of all reporting groups
Arm/Group | IFN-alpha2a 450 Microgram (mcg) | IFN-alpha2a 360 Microgram (mcg) | IFN-alpha2a 270 Microgram (mcg) | IFN-alpha2a 180 Microgram (mcg) | IFN-alpha2a 90 Microgram (mcg) | Total
Number analyzed (Participants) | 3 | 3 | 19 | 26 | 32 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 15 | 19 | 27 | 67
  >=65 years | 0 | 0 | 4 | 7 | 5 | 16
Age, Continuous [Median (Full Range); unit: years] | 47 [25 to 55] | 33 [23 to 65] | 58 [31 to 78] | 54 [35 to 75] | 52 [19 to 78] | 53 [19 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 12 | 17 | 21 | 54
  Male | 1 | 1 | 7 | 9 | 11 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 2 | 3
  White | 3 | 3 | 19 | 23 | 29 | 77
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 19 | 26 | 32 | 83

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete Response (CR) or Partial Response (PR)
Description: CR = Reduction of PLT to <440x109/l and disappearance of thromboembolic events, without the use of anagrelide or hydroxyurea
  PR = Reduction of PLT by 50% but still >440x109/l or reduction of thromboembolic events by 50%, without the use of anagrelide or hydroxyurea
Time Frame: Up to 18 years
Measure: Count of Participants; unit: Participants
Arm/Group | IFN-alpha2a 450 Microgram (mcg) | IFN-alpha2a 360 Microgram (mcg) | IFN-alpha2a 270 Microgram (mcg) | IFN-alpha2a 180 Microgram (mcg) | IFN-alpha2a 90 Microgram (mcg)
Number analyzed (Participants) | 3 | 3 | 19 | 26 | 32
Participants | 3 | 3 | 14 | 23 | 23

ADVERSE EVENTS:
Time Frame: Up to 18 years, one month and 23 days
Arm/Group | IFN-alpha2a 450 Microgram (mcg) | IFN-alpha2a 360 Microgram (mcg) | IFN-alpha2a 270 Microgram (mcg) | IFN-alpha2a 180 Microgram (mcg) | IFN-alpha2a 90 Microgram (mcg)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/19 | 2/26 | 1/32
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 3/19 | 3/26 | 7/32
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 9/19 | 8/26 | 7/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IFN-alpha2a 450 Microgram (mcg) (N=3) | IFN-alpha2a 360 Microgram (mcg) (N=3) | IFN-alpha2a 270 Microgram (mcg) (N=19) | IFN-alpha2a 180 Microgram (mcg) (N=26) | IFN-alpha2a 90 Microgram (mcg) (N=32)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic Aneurism (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
carcinoma-facial (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Condition (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatal Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive adenocarcinoma of the colon (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leg wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgery for post- menopausal bleeding (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Resection of Small Intestine (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IFN-alpha2a 450 Microgram (mcg) (N=3) | IFN-alpha2a 360 Microgram (mcg) (N=3) | IFN-alpha2a 270 Microgram (mcg) (N=19) | IFN-alpha2a 180 Microgram (mcg) (N=26) | IFN-alpha2a 90 Microgram (mcg) (N=32)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 6 (6) | 4 (4) | 2 (2)
Elevated transaminase (Investigations) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blur Vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT00452023/Prot_SAP_000.pdf